CLINICAL TRIAL: NCT00131755
Title: Efficacy of 6 Months Treatment With Diazoxide at Bedtime in Preventing Beta-cell Demise in Newly Diagnosed Type 1 Diabetes
Brief Title: Efficacy of Diazoxide in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grill, Valdemar, M.D. (Individual)
Responsible Party: Valdemar Grill, NTNU
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIAZ 1; Eudract 2004-004103-38
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; beta cell rest; diazoxide; insulin secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diazoxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: diazoxide

SUMMARY:
The purpose of this study is to find out if Diazoxide can partly retain insulin production in newly diagnosed type 1 diabetes patients.

DETAILED DESCRIPTION:
At the time of diagnosis most subjects with type 1 diabetes retain significant endogenous insulin secretion as assessed by C-peptide measurements. Although not sufficient for the needs of the individual, residual insulin secretion is important for metabolic control, for avoidance of hypoglycemic episodes and, perhaps, for protection against diabetic complications. To retain residual endogenous insulin secretion in type 1 diabetes is thus highly desirable.

Residual insulin secretion deteriorates during the course of type 1 diabetes. The underlying autoimmune process is a major determinant of deterioration.

However, also measures that do not directly target the immune system could be beneficial. The DCCT study randomised subjects with type 1 diabetes to either intensive or conventional insulin treatment. The intensive insulin treatment markedly retarded deterioration in C-peptide levels during 5 years of observation. The favourable effect could be due to lesser hyperglycemia per se. Alternatively, the effect of intensive insulin treatment could be secondary to lesser degree of over-stimulation of the patients' beta-cells.

It is by now established that relief from over-stimulation by diazoxide favourably affects beta-cell function and that such treatment can retard a decline in residual insulin secretion in subjects with newly diagnosed type 1 diabetes. Diazoxide has been used in clinical practice for > three decades without major safety concerns.

Disturbing, albeit reversible, side effects are halting long-term studies with diazoxide in type 1 diabetes. The researchers find that lower and intermittent (i.e. night time) dosing of diazoxide produces no measurable side effects in subjects with type 2 diabetes.

This is a double blinded placebo controlled study, with 35 participants with newly diagnosed type 1 diabetes are randomised into either placebo or Diazoxide for 6 months. The patients will be followed up after intervention for at least 12 months.

Beta cell function and glycemic control will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes no longer than three months
* Positive antibodies against GAD or IA2
* Age between 18-40 years
* C-peptide >0.2 nmol/l

Exclusion Criteria:

* Drug or alcohol abuse
* Severe concomitant disease
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Insulin secretion (measured by fasting and stimulated c-peptide) | 12 months
Glycemic control (measured by blood glucose) | 12 months

SECONDARY OUTCOMES:
Autoimmune activity (measured by islet antibodies) | 6 months
Side effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Grill Valdemar, MD PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- University Hospital of Trondheim, Trondheim, Norway